CLINICAL TRIAL: NCT05114291
Title: From Micro- to Macro-vessels : Water, Salt, Heart and Kidneys
Acronym: ConcentRatio
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210934; 2021-A01291-40 (Other: France : Ministry of Health)
Record Dates: First submitted 2021-10-22; First posted 2021-11-09 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
Keywords: Hypertension; Aortic stiffness; Fasting urinary osmolarity; Cardiovascular risk
MeSH Terms: conditions — Hypertension | interventions — Hospitalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Explorations are planned as part of the one-day hospitalization — * Clinical parameters : Interrogation, physical examination, morphological data measurements (weight, height, waist circumference, hip circumference) and impedencemetry (body composition).
  * Biological samples : Blood and urine exam, fasting urine sample (urinary osmolarity)
  * Standardized blood pressure measurement :
    * After 5 to 10 minutes of rest, with automated measurements at 1 minute intervals : "un-attended", then "attended"
  * Hemodynamic parameters :
    * Sphygmocor® : measure of the central blood pressure and pulse wave velocity
    * MESI® tool : measure of the Systolic Pressure Index (PSI or IPS)
    * pOpmetre® : Calculation of the speed of the pulse wave by the pOpmetre® device
  * Others : if indicated (echocardiography, ABPM)

SUMMARY:
Hypertension is a public health concern and affects nearly a third of the French population. It can be complicated by visceral impact (including brain, heart and kidney complications) as well as on vessels especially large arteries, responsible for arterial stiffening. There are close interactions between heart and kidneys, as well as between large arteries and micro-vessels. These relationships also involve the water and salt balance and its regulatory mechanisms. Urinary concentration abilities are closely linked to the renal medullary blood flow, which in itself depends on the integrity of renal micro vessels, thus influencing the water and salt balance. Few previous studies evaluated the interconnections between renal urinary concentration abilities and blood pressure. A previous-one reported a positive relation between pulse pressure and urinary concentration in men, suggesting that subjects with higher urinary osmolarity could present a higher cardiovascular risk. Carotid-femoral pulse wave velocity represents the gold standard for non-invasive arterial stiffness assessment and constitutes an arteriosclerosis infra-clinical marker recommended by the European Society of Cardiology- European Society of Hypertension. It is considered as an independent predictor for global and cardiovascular mortality, coronary heart disease and fatal stroke among patients with hypertension, diabetes or end stage kidney disease. The purpose of this study is to evaluate the relations between fasting urinary osmolarity and arterial stiffness assessed by carotid-femoral pulse wave velocity (CF-PWV) among patients with hypertension.

DETAILED DESCRIPTION:
1. Hypertension

   1. Hypertension, kidneys et urinary sodium excretion

      Kidneys are heavily involved in blood pressure regulation in particular through water and salt balance control, and their impact on vasomotor tone through the renin-angiotensin aldosterone system (RAAS), prostaglandins or atrial natriuretic factor (FAN) actions. They take a central place in blood pressure regulation and indirectly in arterial stiffening.

      Daily urinary sodium excretion represents a major determinant of blood pressure. It is defined as the product of urinary sodium concentration and urinary output. In a steady state, it equals sodium intake. When kidneys are unable to excrete sodium, blood volume and blood pressure increase. The result is an adaptive decrease in sodium reabsorption (called "pressure natriuresis"), in order to restore the sodium balance. "Salt sensitivity" has been defined as a significant increase in blood pressure associated with the increase sodium intake. It has been associated with age, ethnicity, obesity, metabolic syndrome, and chronic kidney disease (CKD). Chronic kidney disease is frequently associated with salt and fluid retention, which promote hypertension and increase cardiovascular risk.

      Among dialysis patients, fluid overload has been widely described as an independent mortality risk factor. Recently, Faucon et al. reported in the nephroTEST cohort of CKD patients not yet on dialysis that the measured extra cellular volume (ECV) was an independent risk factor for mortality but also for CKD progression to the end stage of kidney disease. Reduced sodium excretion abilities associated with CKD progression lead to fluid overload and cardiac consequences. The increase of left ventricular preload promotes diastolic dysfunction. In parallel, the prolonged increase of left ventricular afterload promotes left ventricular hypertrophy. Other CKD associated factors could also contribute to left ventricular hypertrophy such as the increased arterial stiffness, and CKD-mineral and bone disorders including the raise of FGF-23.
   2. Nephron, water and salt balance regulation, and outside of the glomerulus

      The nephron represents the kidney functional unit. It plays a major role in water and salt balance control. "Kidney function" assessment is often reduced to its glomerular functions, including glomerular filtration rate (GFR) and albuminuria level. The other segments of the nephron are however largely involved in this balance control. Their function can be altered even without glomerular dysfunction and therefore without renal insufficiency. Thus, tubular segments, peritubular capillaries and the interstitial space can also be altered in some kidney diseases. These structures, and more particularly the ascending limb of the loop of Henle, the peritubular micro-vessels and the collecting duct, are involved in the corticopapillary gradient creation and maintenance. This gradient is essential for the urine concentrating mechanism. Tubular damages assessed on renal pathology would also be more correlated to impaired urine concentration and acidification than to glomeruli involvement. Fasting urinary osmolarity is a simple, non-invasive marker for assessing urinary concentration abilities. It is yet poorly studied in clinical research. At same level of GFR, its level would be associated with tubular dysfunctions and peritubular vascular lesions, namely with medullary functions. Fasting urinary osmolarity has also been associated with GFR decline and progression of CKD to end stage kidney disease. On the other hand, some of the tubular segments constitute direct targets of systemic hormonal regulation. Aldosterone thus promotes sodium retention and potassium excretion through the activation of mineralocorticoid receptors located on distal tubular cells and the involvement of ENaC and ROMK channels.
   3. Hypertension and urinary concentration

   Perrucca et al. suggested that urinary concentration and its regulatory hormone, antidiuretic hormone (ADH), may contribute to cardiovascular disease susceptibility. ADH binding to its V2R receptor promotes distal reabsorption of free water and thus favors urinary concentration. This hormone has thus an action through kidneys promoting urinary concentration through free water reabsorption, but also a vascular effect leading to vasoconstriction. Hypertension has been associated with increased plasma ADH levels. Zhang et al. thus reported in a cohort of 534 middle-aged subjects, the significant association between plasma ADH levels and blood pressure levels as well as with hypertension, especially in patients with low plasma renin activity. The antidiuretic hormone would also be at higher levels in men than in women, as well as in African American subjects compared to Caucasians, likewise hypertension is also more frequent in these two populations.

   Furthermore, Bankir et al. described in a retrospective cohort of 141 healthy subjects of 18 to 40 years old that black individuals presented significantly higher urine concentration and lower urinary volume than white individuals. In addition, a significant and positive relationship between urinary concentration levels and pulse pressure was found among men. This association was more marked among black individuals compared to white individuals. Since pulse pressure is currently considered as an independent risk factor for cardiovascular disease, associated with both cardiovascular morbidity (increased incidence of myocardial infarction or congestive heart failure) and cardiovascular mortality from coronary artery disease, an association between urinary concentration abilities and cardiovascular risk could be considered. In addition, urine dilution by increasing water intake is one of the main objective in the management of lithiasis patients. The increase of urinary concentration is indeed associated with an increased risk of crystallization and therefore an increased risk of kidney stones recurrence. Lithiasis patients have also been described as a population with an increased cardiovascular risk. These additional elements support the hypothesis of a potential association between urinary concentration and cardiovascular risk.
2. Arterial stiffness

   1. Hypertension, arteriosclerosis and evaluation

      Arteriosclerosis represents an arterial degeneration process associated with physiological aging but much more marked in some pathological circumstances such as hypertension, diabetes or chronic kidney disease. The arterial wall involvement concerns the media of large arteries, unlike atherosclerosis in which the involvement initially involves the intima, resulting in an accelerated stiffening of the vascular tree. Large arteries stiffening can induce myocardial hypertrophy, favors heart failure, arrhythmias and even myocardial ischemia. Carotid-femoral pulse wave velocity enables non-invasive assessment of central arterial stiffness. It currently represents the gold standard for non-invasive arterial stiffness measurements and constitutes an arteriosclerosis infra-clinical marker recommended by the European Society of Cardiology- European Society of Hypertension. In practice, it corresponds to the velocity at which the pulse wave propagates over a specific arterial segment. The pulse wave travels slowly through flexible and elastic arteries, and rapidly through rigid arteries. CF-PWV measurement requires an automated software. It is a simple, non-invasive, validated, robust, reproducible and accessible procedure in clinical practice.
   2. Arterial stiffness and cardiovascular risk

      CF-PWV thus enables us to detect large arteries damages at an infra-clinical stage and to identify populations at high cardiovascular risk. It has been described as an independent predictor for global and cardiovascular mortality, coronary heart disease and fatal stroke in many populations: in the general population, in elderly patients, in patients with diabetes, with hypertension, in CKD-patients, patients with end-stage kidney disease, and also in renal transplant recipients. Aortic stiffness has been shown to be predictive of cardiovascular events, independently and beyond traditional risk factors and the Framingham score.
   3. Arterial stiffness and fluid overload

      Fluid overload can also contribute to structural and functional alterations in large arteries and therefore promote arterial stiffness. The increase in venous pressure induced by sodium overload initiates a vicious circle. The result is an increase in renal interstitial pressure, which disrupts renal blood flow, and promotes further retention. Plasma volume expands, increasing venous pressure further. The associated increase in filling pressures could thus promote structural and functional alteration of large arteries.

      Furthermore, the diastolic blood pressure decrease induce a reduction in coronary perfusion pressure, which contributes to myocardial ischemia. In case of heart failure, sodium retention is associated with a defective arterial filling. Urinary sodium excretion decreases while sodium and fluid overload increases.
   4. Micro- and macro-vessels relationships

   Safar et al. previously reported the links between macro- and micro-vessels evidenced by mouse models of hypertension and human studies. Indeed, pulse pressure increase associated with arterial compliance disturbances promotes impaired microcirculation, particularly in kidneys. An alteration of the extracellular matrix could involve both vascular smooth muscle cells (VSMCs) and renal cells. Several underlying physiopathological mechanisms have been suggested, involving notably the water and salt balance and the hormonal systemic regulatory mechanisms including the renin-angiotensin-aldosterone system. Urinary concentration abilities are closely linked to the renal medullary blood flow which itself depends on the renal microcirculation integrity.
3. Studied-population

This study focus on patients with severe/resistant hypertension and/or with suspicion of secondary hypertension, who are addressed in a one-day hospitalization to benefit from standardized examinations including hormonal analyses (renin - aldosterone ± plasma cortisol). These hypertensive patients present an increased cardiovascular risk. The CF-PWV measure enables aortic stiffness assessment. It constitutes an arteriosclerosis infra-clinical marker recommended by the European Society of Cardiology- European Society of Hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients
* Day hospitalization for a check-up in the context of arterial hypertension with suspicion of secondary origin including a dosage of renin and plasma aldosterone
* Non-opposition to the study

Exclusion Criteria:

* Cardiac arrythmia
* Patient under AME (state medical assistance)
* Treatments interfering with uninterrupted hormonal dosages before day hospitalization

  * Absence of B-blockers, converting enzyme inhibitor and sartans in the 15 days preceding the dosages
  * Absence of antialdosterone, and amiloride in the 6 weeks preceding the dosages
  * Absence of loop diuretics or diuretics in the 7 days preceding the dosages

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study concerns patients with hypertension who are addressed to a one-day hospitalization in order to realize standardized examinations (must include hormonal analyses : renin and aldosterone)
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
CF-PWV | Inclusion
  Carotid-femoral pulse wave velocity

SECONDARY OUTCOMES:
PRA | Inclusion
  Plasma renin activity
Nocturnal dipping percentage of systolic blood pressure | Inclusion
  Nocturnal dipping percentage of systolic blood pressure
Smoking status | Inclusion
  Declared smoking status
Ankle-brachial pressure index (ABPI) | Inclusion
  Ankle-brachial pressure index (ABPI)
Primary hyperaldosteronism | Inclusion
  Primary hyperaldosteronism diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Lynda CHEDDANI, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Centre Interdisciplinaire de Thérapeutique et d'Education APHP- Hôtel Dieu Hospital, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No